CLINICAL TRIAL: NCT00846235
Title: Clinical Evaluation of the Effect of Moisturising Cream on Skin Moisture in Atopic Dermatitis
Brief Title: Effect of Moisturising Creams on Skin Moisture in Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Kimmo Ingman MD PhD, Orion Corporation, Orion Pharma, R&D
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2934004
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis; Atopic; Moisturising cream; Skin
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moisturising cream (Experimental)
  Interventions: Other: Aqualan L, Aqualan Plus, Aqualan L + glycerol ad 20%

INTERVENTIONS:
Other: Aqualan L, Aqualan Plus, Aqualan L + glycerol ad 20% — moisturising cream twice daily three weeks

SUMMARY:
The aim of this study is evaluate the effect of three moisturising creams on Stratum corneum (SC) hydratation and barrier function.

DETAILED DESCRIPTION:
In the present study, 24 subjects with AD will be treated for 3 weeks twice daily by using 3 different moisturising creams. Duration of the study is based on literature. Various moisturising creams containing glycerol have been reported to be beneficial for AD lesions. The optimal glycerol content in moisturising creams is not known. The secondary objective is the comparison of change in the SC water content and in the TEWL from the skin surface from the baseline to the end of study between different moisturizing creams containing different amount of glycerol.

Change in the SC water content and in the TEWL can be demonstrated with noninvasive instrumental measurement. The treated skin will be followed up instrumentally, and one measurement area will serve as an untreated control. The primary evaluation is the comparison of change in the SC water content and in the TEWL on the skin surface from the baseline to the end of study between the 4 treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (IC) obtained.
2. 18-55 years of age, Caucasian, Finnish speaking, male or female subjects.
3. Weight at least 50 kg.
4. Body mass index (BMI) 18-30 kg/m2.
5. Clinical assessment for the diagnosis of mild or moderate atopic dermatitis

Exclusion Criteria:

1. Any clinically relevant medical condition judged by the investigator.
2. Any known allergy to ingredients of the test treatments.
3. Any systemic immunosuppressive or cortisone medication.
4. UV-Light therapy and sunlight exposure within 30 days prior to the start of the study and during study.
5. Any abnormal physical finding which may interfere with the interpretation of test results or cause a health risk for the subject if he/she participates in the study.
6. Anticipated difficulty related to stopping of caffeine intake during study centre visits.
7. Current use of nicotine containing products more than 5 cigarettes (or equivalent)/day and inability to refrain from the use of nicotine containing products during the study.
8. Recent or current drug abuse or suspected abuse or positive result in screening of drug abuse.
9. Recent or current alcohol abuse (more than 16 units/week for women and more than 21 units/week for men) or suspected abuse.
10. Participation in another clinical study within 30 days prior to the start of the present study.
11. Predictable poor compliance or inability to communicate well with the investigator.
12. Inability to participate in all treatment periods.
13. Pregnant or lactating females.
14. Females of childbearing potential if they are not using proper contraception (hormonal contraception, intrauterine device (IUD) or surgical sterilization, spermicidal foam in conjunction with condom on male partner) (Note: women of childbearing potential with no current sexual relationship can be included without contraception according to the judgement of the investigator).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Skin hydratation and transepidermal water loss. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nykänen, PhD, Study Director — Orion Pharma, R&D, Translational Sciences, Finland
Locations (1):
- Orion Pharma R&D, Espoo, Finland